CLINICAL TRIAL: NCT04161443
Title: Effect of Quadratus Lumborum Muscle Energy Technique Along With Gluteus Medius Strengthening Verus Gluteus Medius Strengthening Alone in the Management of Sacroilliac Joint Dysfunction.; A Randomized Controlled Trial.
Brief Title: Effect of Quadratus Lumborum Muscle Energy Technique in Sacroilliac Joint Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Rabail Soomro, Dr. Rabail Rani Soomro, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 019
Record Dates: First submitted 2019-10-30; First posted 2019-11-13 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Sacroiliac Disorder
Keywords: MET, Quadratus lumborum, Sacroilliac joint
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding will be used as the subjects and the assessor both will be blinded for the treatment used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Following physiotherapy treatment will be given to the participants in this group for 4 weeks and each session last for 30 minutes.
  i. MET Quadratus lumborum ii. Ultrasound iii. Gluteus medius exercises iv. Hamstring stretch Posture advice and home exercise program
  Interventions: Other: physiotherapy
- Comparator (Active Comparator): Following physiotherapy treatment will be given to the participants in this group for 4 weeks and each session last for 30 minutes.
  i. Ultrasound ii.Gluteus medius exercises iii.Hamstring stretch
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — * Treatment will be performed three sessions per week for 4 weeks with postural advice and home exercise program with daily record of home diary.
  * The selected outcome measures will be taken on initial visit (pre intervention), session 6 and final session 12 (post intervention).

SUMMARY:
Sacroiliac joint as a potential source of low back pain is an overlooked problem. Yet, in the existing years there has been an increasing interest in sacroiliac joint as a pain originator and more attention is being paid into its assessment and treatment in the current literature. Muscle imbalance due to postural dysfunction involves mainly gluteus medius and hamstring; however the role of quadratus lumborum working on compensatory mechanism and its treatment effect in the management of sacroiliac joint dysfunction is yet not discovered.

DETAILED DESCRIPTION:
Going through current literature, it is evident that sacroiliac joint dysfunction as a postural dysfunction is highly prevalent among adult population. This dysfunction due to major muscle imbalances if not treated timely can result in serious consequences later in life where it becomes the permanent dysfunction involving the major changes in the joint itself. Muscle imbalance due to postural dysfunction involves mainly gluteus medius and hamstring; however the role of quadratus lumborum working on compensatory mechanism and its treatment effect in the management of sacroiliac joint dysfunction is yet not discovered. All patients will be assessed and screened by consultants as indicated and will refer to physiotherapy with diagnosed non- specific chronic back pain.Patients will further be screened for SIJ dysfunction by physiotherapist.Only those patients who fulfill the criteria of Quadratus lumborum tightness & Gulteus medius weakness will randomly be selected and the sample of 70 will finally be selected for intervention.Written consent form will be taken from all study participants.Simple randomization technique will be used through "Randomization Main" software and randomization sheet will be generated. Patients will be further be assigned equally into two groups as per randomization sheet.Treatment will be performed three sessions per week for 4 weeks with postural advice and home exercise program with daily record of home diary. The selected outcome measures will be taken on initial visit (pre intervention), session 6 and final session 12 (post intervention).

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with unilateral non-specific LBP

  * The Subjects having at least 3 pain provocative tests of SIJ positive out of 5.
  * Age 30-50 years. Both male and female.
  * Pain history greater than six weeks.
  * SIJ diagnostic scoring cut off point 4.
  * VAS cut off point mild to moderate.

Exclusion Criteria:

* Radiating pain with sensory or motor deﬁcits.
* History of fracture or any spinal surgery
* Trauma
* Any dysfunction of hip or knee
* Any systemic disease.
* Pregnancy

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
visual analog scale to measure the change in level of Pain intensity | Total duration of treatment is 4 weeks and 12 sessions, 3 sessions per week on alternate days. Patients will be assessed at baseline, at 6th session at the end of 2nd week and 12th session at the end of 4th week.
  A Visual Analogue ScalE is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end ranging from no pain to severe pain.
Oswestry Disability Index to measure change in level of disability | Total duration of treatment is 4 weeks and 12 sessions, 3 sessions per week on alternate days. Patients will be assessed at baseline, at 6th session at the end of 2nd week and 12th session at the end of 4th week.
  Change in level of disability as evaluated by means of Oswestry Disability Index 2.0 (ODI)
SF-36 QUALITY OF LIFE to measure change in general health | Total duration of treatment is 4 weeks and 12 sessions, 3 sessions per week on alternate days. Patients will be assessed at baseline and 12th session at the end of 4th week.
  SF-36 measure 8 different health concepts including general health, physical functioning, role functioning, bodily pain, mental health, emotional functioning, vitality, and social functioning.

SECONDARY OUTCOMES:
Hand Held Dynamometer to check gluteus medius muscle strength | Total duration of treatment is 4 weeks and 12 sessions, 3 sessions per week on alternate days. Patients will be assessed at baseline, at 6th session at the end of 2nd week and 12th session at the end of 4th week.
  The strength of the gluteus medius muscle was assessed on the dominant side using the Microfet2 hand-held dynamometer (MicroFET 2, Hoogan Health Industries, West Jordan, UT, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Rabail Soomro, Principal Investigator — University of Lahore; Hussain Kari mi, Study Chair — University of Lahore
Locations (1):
- Institute of physical medicine and rehabilitation, Dow University of health sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No